CLINICAL TRIAL: NCT04480996
Title: Evaluation of Reporting of Road Traffic Accidents With Drugs Responsible for Cognitive and Psychomotor Side Effects (ERoADS)
Brief Title: Evaluation of Reporting of Road Traffic Accidents With Drugs Responsible for Cognitive Side Effects (ERoADS)
Acronym: ERoADS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20200619
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-06

CONDITIONS: Accident, Traffic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Road traffic accidents with medicines: Road traffic accidents cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of patients treated by Drugs Responsible for Cognitive and Psychomotor Side Effects
  Interventions: Drug: Drugs Responsible for Cognitive Side Effects

INTERVENTIONS:
Drug: Drugs Responsible for Cognitive Side Effects — identification of road traffic accidents associated with drugs responsible for psychomotor side effects
  Other Names: Drugs Responsible for Pyschomotor Side Effects

SUMMARY:
Drugs responsible for cognitive and psychomotor side effects may lead to impaired driving skills and road traffic accidents. This study investigates reports of road traffic accident for different class of drugs responsible for cognitive and psychomotor sides effects (pyschotropic agents, neurotropic agents, antineoplasic agents) in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
Some medications are responsible of a wide range of cognitive and psychomotor side effects that may make it unsafe to drive and lead to risks of road accidents .The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of road traffic accidents following treatment with different class of drugs responsible for pyschomotor sides effects.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/03/2020
* Adverse events reported were including the MedDRA terms: Road Traffic Accident (SMQ)
* Patients treated with at least one liable nervous system drugs (ATC class N) or that can induce cognitive and pyschomotor undesirable effects by crossing the blood-brain barrier (ATC class A04, C02A, L)

Exclusion Criteria:

* Chronology not compatible between the drug and the road traffic accident

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated With Drugs Responsible for Cognitive and Psychomotor Side Effects
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Association between drugs responsible for cognitive and psychomotor side effects and road traffic accidents cases | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2020
  Identification of cases with association between each individual of different class of drugs responsible for cognitive ans psychomotor side effects and road traffic accidents cases

SECONDARY OUTCOMES:
Association between two drugs of the same class, leading to an over-reporting of road traffic accidents | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2020
  Association between two drugs in the different class studied and road traffic accidents cases to search for a potential interaction between two drugs of the same class, leading to an over-reporting of road traffic accidents
Description of the population of patients having a road traffic accident related to taking medication | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2020
  Identification of the population criteria (age, sex ...) having road accidents related to certain classes of drugs

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Lelong-Boulouard, PhD, PharmD, Principal Investigator — CHU CAEN
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

REFERENCES:
- [Derived] Chretien B, Nguyen S, Dolladille C, Morice PM, Heraudeau M, Loilier M, Fedrizzi S, Bourgine J, Cesbron A, Alexandre J, Bocca ML, Freret T, Lelong-Boulouard V. Association between road traffic accidents and drugs belonging to the antiseizure medications class: A pharmacovigilance analysis in VigiBase. Br J Clin Pharmacol. 2023 Jan;89(1):222-231. doi: 10.1111/bcp.15481. Epub 2022 Aug 21. PMID 35939367